CLINICAL TRIAL: NCT02369796
Title: An Open-Label, Phase 2a Study to Evaluate the Pharmacodynamics of Different Dosing Regimens of TAK-448, a Kisspeptin Agonist, in Male Overweight/Obese Participants With Hypogonadotropic Hypogonadism
Brief Title: A Phase 2a Pharmacodynamic Study of TAK-448 in Participants With Hypogonadotropic Hypogonadism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate the study because the study did not achieve the primary efficacy objective.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-448-2001; U1111-1162-4892 (Registry Identifier: WHO); 2014-002155-25 (EudraCT Number); 14/LO/1950 (Registry Identifier: NRES)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Hypogonadotropic Hypogonadism
Keywords: Drug therapy
MeSH Terms: conditions — Hypogonadism | interventions — metastin (46-54), acetyl-tyrosyl(46)-hydroxypropyl(47)-threonyl(49)-azaglycyl(51)-methylarginyl(53)-tryptophyl(54)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- TAK-448 3 µg once weekly (Experimental): TAK-448 3 µg, subcutaneous injection, once weekly on Days 1, 8, 15 and 22.
  Interventions: Drug: TAK-448
- TAK-448 1 µg once weekly (Experimental): TAK-448 1 µg, subcutaneous injection, once weekly on Days 1, 8, 15 and 22.
  Interventions: Drug: TAK-448
- TAK-448 0.3 µg once weekly (Experimental): TAK-448 0.3 µg, subcutaneous injection, once weekly on Days 1, 8, 15 and 22.
  Interventions: Drug: TAK-448
- TAK-448 0.3 µg twice weekly (Experimental): TAK-448 0.3 µg, subcutaneous injection, twice weekly on Days 1, 4, 8, 11, 15, 18, 22, and 25.
  Interventions: Drug: TAK-448
- TAK-448 0.1 µg twice weekly (Experimental): TAK-448 0.1 µg, subcutaneous injection, twice weekly on Days 1, 4, 8, 11, 15, 18, 22, and 25.
  Interventions: Drug: TAK-448

INTERVENTIONS:
Drug: TAK-448 — TAK-448 solution for subcutaneous injection

SUMMARY:
The purpose of this study is to evaluate the effects on serum testosterone after 4 weeks of subcutaneous (SC) dose administration, with different doses and dosing frequencies of TAK-448 to overweight/obese males with hypogonadotropic hypogonadism.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-448. TAK-448 is being tested to treat overweight/obese males with hypogonadotropic hypogonadism. This study will look at the effects of TAK-448 on serum testosterone at different doses and different dosing frequencies.

The study will enroll 15 patients. There will be 5 cohorts and participants will be assigned to cohorts in sequential order. Cohorts will be assigned to the following treatment groups:

* TAK-448 3 µg once weekly
* TAK-448 1 µg once weekly
* TAK-448 0.3 µg once weekly
* TAK-448 0.3 µg twice weekly
* TAK-448 0.1 µg twice weekly

All participants will be administered study drug via SC injection once or twice a week depending on their assigned cohort for four weeks.

This single-center trial will be conducted in the United Kingdom. The overall time to participate in this study is up to 32 days. Participants will make multiple visits to the clinic (depending once-weekly or twice-weekly dosing), and will be contacted by telephone 1 week after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant has two morning total serum testosterone (ST) concentrations ≤12.0 nmol/L (≤3.46 ng/mL) taken during the Screening period.
4. Is male and aged 18 to 60 years, inclusive.
5. Has a body mass index (BMI) between 25.0 and 50.0 kg/m^2, inclusive.
6. If diagnosed with type II diabetes mellitus (T2DM), has a glycosylated hemoglobin (HbA1c) concentration <12% at Screening and is on a stable dose of up to 4 diabetes therapies (including insulin and/or glucagon-like peptide-1 therapies).
7. Has a luteinizing hormone (LH) concentration <8 IU/L at Screening.
8. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening.
2. Has received TAK-448 in a previous clinical study, or previous cohort.
3. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality (other than T2DM, its complications and associated conditions), which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a recent history or clinical manifestations of significant cardiovascular disease (CVD) - such as a history of myocardial infarction or stroke in the 6 months preceding the Screening visit or has untreated peripheral arterial disease.
6. Has a history of hypersensitivity or allergies to any component of the formulation of TAK-448.
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 5 years prior to Screening.
8. Is required to take excluded medications, supplements, or food products.
9. Intends to donate sperm during the course of this study or for 12 weeks after the last dose of study drug.
10. Has clinical evidence of anatomic or pathological hypothalamic/pituitary disease.
11. Is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking TAK-448, or a similar drug in the same class that might interfere with the conduct of the study.
12. Has a history of cancer (including prostate cancer), with the exception of basal cell carcinoma which has been in remission for at least 5 years prior to Screening.
13. Has a history of or present prostate disease (including benign prostatic hyperplasia) or prostate-specific antigen (PSA) is >4 ng/mL at Screening.
14. Has a known history of human immunodeficiency virus infection at Screening.
15. Is deemed by the study team to have poor peripheral venous access.
16. Has donated or lost 450 mL or more of his blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days prior to Screening, or is planning to donate blood for 12 weeks after the last dose of study medication.
17. Has a Screening or Day -1 abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature of the principal investigator or medically qualified subinvestigator.
18. Has abnormal Screening or Day -1 laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2× the upper limits of normal (ULN).
19. The participant, in the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.
20. Has had more than two severe hypoglycemic events (requiring third party assistance) within 6 months prior to the Screening Visit.
21. Has a diagnosis of type 1 diabetes mellitus.
22. Has a history of diabetic ketoacidosis.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Oxford, Oxfordshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United Kingdom from 10 February 2015 to 3 November 2015.
Pre-assignment Details: Overweight/obese male participants with a diagnosis of hypogonadotropic hypogonadism were enrolled in 1 of 5 treatment groups: once weekly TAK-448 3 µg, 1 µg or 0.3 µg or twice weekly TAK-448 0.3 µg or 0.1 µg.
Period: Overall Study
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly | TAK-448 0.3 µg Twice Weekly | TAK-448 0.1 µg Twice Weekly
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were enrolled and received at least 1 dose of study drug, including participants who did not complete all scheduled study visits.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly | TAK-448 0.3 µg Twice Weekly | TAK-448 0.1 µg Twice Weekly | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (8.02) | 50.7 (4.62) | 51.7 (3.79) | 56.0 (3.61) | 45.0 (19.16) | 50.8 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 3 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 0 | 0 | 0 | 0 | 2
  White | 1 | 3 | 3 | 3 | 3 | 13
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 | 3 | 3 | 3 | 3 | 15
Height [Mean (Standard Deviation); unit: cm] | 168 (7) | 174 (6) | 181 (18) | 178 (6) | 178 (12) | 176 (10)
Weight [Mean (Standard Deviation); unit: kg] | 104 (30) | 113 (10) | 119 (26) | 115 (7) | 110 (26) | 112 (19)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 36 (8) | 37 (1) | 36 (2) | 36 (2) | 34 (4) | 36 (4)
Smoking Classification [Number; unit: participants]
  Has never smoked | 3 | 0 | 0 | 1 | 1 | 5
  Is current smoker | 0 | 0 | 1 | 0 | 0 | 1
  Is an ex-smoker | 0 | 3 | 2 | 2 | 2 | 9
Alcohol Classification [Number; unit: participants]
  Has never drunk | 0 | 0 | 1 | 0 | 0 | 1
  Is current drinker | 3 | 2 | 1 | 2 | 2 | 10
  Is an ex-drinker | 0 | 1 | 1 | 1 | 1 | 4
Caffeine Consumption [Number; unit: participants]
  Yes | 3 | 3 | 3 | 2 | 3 | 14
  No | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Mean Area Under the Effect Curve From Time 0 to 72 Hours (AUEC72) of Total Serum Testosterone for Once Weekly Dosing Groups
Description: Area under the pharmacodynamic (PD) total serum testosterone (ST) concentration-time curve from the time 0 to 72 hours, calculated using the linear trapezoidal rule for baseline profile and those obtained after first and last dose.
Time Frame: Baseline and Day 22 pre-dose and multiple time points (up to 72 hours) post dose
Population: PD set included all participants who received at least one dose of study drug and had at least 1 valid PD measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly
Number analyzed (Participants) | 3 | 3 | 3
percent change | 1.9 (11.3) | 13.5 (24.9) | 14.9 (16.3)

2. Primary Outcome: Percent Change From Baseline in Mean Area Under the Effect Curve From Time 0 to 72 Hours (AUEC72) of Total Serum Testosterone for Twice Weekly Dosing Groups
Description: Area under the PD total ST concentration-time curve from the time 0 to 72 hours, calculated using the linear trapezoidal rule for baseline profile and those obtained after first and last dose.
Time Frame: Baseline and Day 25 pre-dose and multiple time points (up to 72 hours) post dose
Population: PD set included all participants who received at least one dose of study drug and had at least 1 valid PD measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-448 0.3 µg Twice Weekly | TAK-448 0.1 µg Twice Weekly
Number analyzed (Participants) | 3 | 3
percent change | -2.8 (3.7) | 6.0 (12.3)

3. Primary Outcome: Percent Change From Baseline in Mean Area Under the Effect Curve From Time 0 to 72 Hours (AUEC72) of Free Serum Testosterone for Once Weekly Dosing Groups
Description: Area under the PD free ST concentration-time curve from the time 0 to 72 hours, calculated using the linear trapezoidal rule for baseline profile and those obtained after first and last dose.
Time Frame: Baseline and Day 22 pre-dose and multiple time points (up to 72 hours) post dose
Population: PD set included all participants who received at least one dose of study drug and had at least 1 valid PD measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly
Number analyzed (Participants) | 3 | 3 | 3
percent change | 3.55 (9.08) | 11.1 (28.0) | 7.92 (8.88)

4. Primary Outcome: Percent Change From Baseline in Mean Area Under the Effect Curve From Time 0 to 72 Hours (AUEC72) of Free Serum Testosterone for Twice Weekly Dosing Groups
Description: as for outcome 3
Time Frame: Baseline and Day 25 pre-dose and multiple time points (up to 72 hours) post dose
Population: PD set included all participants who received at least one dose of study drug and had at least 1 valid PD measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-448 0.3 µg Twice Weekly | TAK-448 0.1 µg Twice Weekly
Number analyzed (Participants) | 3 | 3
percent change | -9.00 (4.23) | 20.5 (5.33)

5. Primary Outcome: Trough Serum Concentration (Ctrough) of Total Serum Testosterone for Once Weekly Dosing Groups
Description: Trough serum concentration of total ST, defined as lowest baseline concentration compared to pre-dose of the last dose.
Time Frame: Day 22 pre-dose
Population: PD set included all participants who received at least one dose of study drug and had at least 1 valid PD measure.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly
Number analyzed (Participants) | 3 | 3 | 3
nmol/L | 5.4 (1.3) | 4.4 (3.1) | 8.7 (1.3)

6. Primary Outcome: Trough Serum Concentration (Ctrough) of Total Serum Testosterone for Twice Weekly Dosing Group
Description: Trough serum concentration of total ST, defined as lowest baseline concentration compared to pre-dose of the last dose.
Time Frame: Day 25 pre-dose
Population: PD set included all participants who received at least one dose of study drug and had at least 1 valid PD measure.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | TAK-448 0.3 µg Twice Weekly | TAK-448 0.1 µg Twice Weekly
Number analyzed (Participants) | 3 | 3
nmol/L | 4.7 (2.8) | 6.9 (2.1)

7. Primary Outcome: Trough Serum Concentration (Ctrough) of Free Serum Testosterone for Once Weekly Dosing Groups
Description: Trough serum concentration of free ST, defined as lowest baseline concentration compared to pre-dose of the last dose.
Time Frame: Day 22 pre-dose
Population: PD set included all participants who received at least one dose of study drug and had at least 1 valid PD measure. Number of participants analyzed is number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly
Number analyzed (Participants) | 3 | 3 | 2
nmol/L | 0.16 (0.03) | 0.12 (0.07) | 0.21 (0.004)

8. Primary Outcome: Trough Serum Concentration (Ctrough) of Free Serum Testosterone for Twice Weekly Dosing Groups
Description: Trough serum concentration of free ST, defined as lowest baseline concentration compared to pre-dose of the last dose.
Time Frame: Day 25 pre-dose
Population: PD set included all participants who received at least one dose of study drug and had at least 1 valid PD measure.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | TAK-448 0.3 µg Twice Weekly | TAK-448 0.1 µg Twice Weekly
Number analyzed (Participants) | 3 | 3
nmol/L | 0.12 (0.09) | 0.20 (0.06)

9. Secondary Outcome: Cmax: Mean Maximum Observed Plasma Concentration for TAK-448 Free Base Form (TAK-448F)
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1 and Day 22 pre-dose and at multiple time points (up to 8 hours) post-dose
Population: Pharmacokinetic (PK) set included all participants who received at least one dose of study drug and had at least 1 measurable concentration of TAK-448F.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly
Number analyzed (Participants) | 3 | 3 | 1
pg/mL
  Day 1 | 39.50 (4.943) | 10.46 (1.484) | NA (NA) — Data was not estimable as plasma concentration was below the lower level of quantification (LLOQ).
  Day 22 | 40.10 (6.344) | 12.27 (3.618) | NA (NA) — Data was not estimable as plasma concentration was below LLOQ.

10. Secondary Outcome: AUC(0-∞): Mean Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-448F
Description: AUC(0-∞) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: Day 1 and Day 22 pre-dose and at multiple time points (up to 8 hours) post-dose
Population: PK set included all participants who received at least one dose of study drug and had at least 1 measurable concentration of TAK-448F. Here, 'n' is the participants who were analyzed at specific time point.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly
Number analyzed (Participants) | 3 | 1 | 1
pg*hr/mL
  Day 1 (n=3, 0 1) | 112.00 (5.686) | NA (NA) — No participant was analyzed at this time point. | NA (NA) — Data was not estimable as plasma concentration was below LLOQ.
  Day 22 (n=3, 1, 1) | 122.33 (10.477) | 33.30 (NA) — Only 1 participant was analyzed at this time point. | NA (NA) — Data was not estimable as plasma concentration was below LLOQ.

11. Secondary Outcome: AUC(0-tlqc): Mean Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-448F
Description: AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Time Frame: Day 1 and Day 22 pre-dose and at multiple time points (up to 8 hours) post-dose
Population: PK set included all participants who received at least one dose of study drug and had at least 1 measurable concentration of TAK-448F.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly
Number analyzed (Participants) | 3 | 3 | 1
pg*hr/mL
  Day 1 | 92.23 (6.732) | 19.00 (3.470) | NA (NA) — Data was not estimable as plasma concentration was below LLOQ.
  Day 22 | 95.20 (11.914) | 18.37 (3.069) | NA (NA) — Data was not estimable as plasma concentration was below LLOQ.

12. Secondary Outcome: Mean Terminal Phase Elimination Half-life (T1/2) for TAK-448F
Description: Terminal Phase Elimination Half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Day 1 and Day 22 pre-dose and at multiple time points (up to 8 hours) post-dose
Population: Pharmacokinetic (PK) set included all participants who received at least one dose of study drug and had at least 1 measurable concentration of TAK-448F. Here, 'n' is the participants who were analyzed at specific time point.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly
Number analyzed (Participants) | 3 | 1 | 1
hr
  Day 1 (n=3, 0, 1) | 1.800 (0.0751) | NA (NA) — No participant was analyzed at this time point. | NA (NA) — Data was not estimable as plasma concentration was below LLOQ.
  Day 22 (n=3, 1, 1) | 2.073 (0.1920) | 1.150 (NA) — Only 1 participant was analyzed at this time point. | NA (NA) — Data was not estimable as plasma concentration was below LLOQ.

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 39
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-448 3 µg Once Weekly | TAK-448 1 µg Once Weekly | TAK-448 0.3 µg Once Weekly | TAK-448 0.3 µg Twice Weekly | TAK-448 0.1 µg Twice Weekly
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/3 | 3/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-448 3 µg Once Weekly (N=3) | TAK-448 1 µg Once Weekly (N=3) | TAK-448 0.3 µg Once Weekly (N=3) | TAK-448 0.3 µg Twice Weekly (N=3) | TAK-448 0.1 µg Twice Weekly (N=3)
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.